CLINICAL TRIAL: NCT02653573
Title: myHEART (My Hypertension Education and Reaching Target) Program: a Feasibility Study of a Young Adult Hypertension Intervention
Brief Title: Young Adult Hypertension Feasibility Study
Acronym: myHEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1297
Record Dates: First submitted 2015-12-28; First posted 2016-01-12 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Health Behavior; Hypertension
Keywords: young adult
MeSH Terms: conditions — Health Behavior; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Telephone health coaching over 3 months with supporting education materials.
  Interventions: Behavioral: Coaching

INTERVENTIONS:
Behavioral: Coaching — Self-management education

SUMMARY:
This study was designed to evaluate the feasibility of a telephone-based health coach self-management intervention for young adults.

DETAILED DESCRIPTION:
To address the unmet need for hypertension care in young adults, MyHEART (My Hypertension Education and Reaching Target), a multi-component hypertension intervention was developed. Eligible patients were identified via the healthcare system's electronic health record.

Inclusion criteria included:

1. 18-39 years old at the start of the study,
2. previous hypertension ICD-9 coded office visits and
3. uncontrolled hypertension (≥140/90 mmHg) based on the last ambulatory blood pressure reading.

Exclusion criteria included a pre-defined list of co-morbidities, in addition to planned or current pregnancy, any health condition that limits physical activity or dietary changes, current participation in another study, and planning to leave the area in the next three months. During the feasibility study, all participants continued to receive usual hypertension care from their primary care provider. The intervention involved health coach calls over a 3-month period using self-management modules. The order of the modules was guided by the participant's choice. All encounters were documented in the electronic health record. Patient acceptability and home blood pressure monitoring survey data was acquired.

ELIGIBILITY:
Inclusion Criteria:

* 18-39 years old at the start of the study
* previous hypertension ICD-9 coded office visits
* uncontrolled hypertension (≥140/90 mmHg) based on the last ambulatory blood pressure reading

Exclusion Criteria:

* Chronic Kidney Disease (Stage 4 or 5 or Dialysis)
* Congestive Heart Failure, Any Etiology
* Activated Healthcare Power of Attorney
* Skilled nursing facility or correctional facility residence
* Currently enrolled in case management or chronic disease management support services
* Sensitive condition diagnosis (e.g. HIV)
* Prescribed warfarin, novel oral anticoagulant, or insulin
* Diagnosis of sickle cell anemia or cystic fibrosis
* Prior stroke, myocardial infarction, coronary artery revascularization
* Syncope within past 12 months
* Prior or planned organ transplant
* Chemotherapy or radiation therapy within 6 months
* Severely impaired hearing or speech
* Current participation in another research study
* Pregnant/planning to become pregnant in the next 12 months
* Planning to leave the area in the next 3 months
* Any health condition that will limit physical activity or dietary changes
* Illegal drug use (other than marijuana) in the past 30 days (Self-report)
* Unable to read or communicate in English

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 3 months
  Patient satisfaction survey of feasibility study

SECONDARY OUTCOMES:
Out-of-clinic blood pressures | 3 months
  Frequency of home or out-of-clinic blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Johnson, MD, MS, Principal Investigator — University of WI School of Medicine and Public Health

IPD SHARING:
Plan to Share IPD: Undecided